CLINICAL TRIAL: NCT05891730
Title: A Detailed Exploration of The Perspectives and Experiences of Patients in Colorectal Cancer Clinical Trials
Brief Title: Examination of Trends in Colorectal Cancer Patients' Clinical Study Experiences
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 82251637
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical study participation percentages haven't always been fully representative of a given demographic.

Participation in this observational clinical research is extremely valuable since it allows people with colorectal cancer to contribute their own experiences and unique viewpoints.

These vital contributions have the potential to affect the development of novel therapies and support services dramatically.

Trial's findings will be critical in furthering the understanding of colorectal cancer, ultimately leading to better patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of colorectal cancer
* Patient has self-identified as planning to enroll in a clinical trial for colorectal cancer
* Patient is at least 18 years of age

Exclusion Criteria:

* Inability to perform regular electronic reporting
* Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients who are actively considering involvement in an observational clinical study, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a colorectal cancer clinical study. | 3 months
Number of colorectal cancer patients who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Winkels RM, Heine-Broring RC, van Zutphen M, van Harten-Gerritsen S, Kok DE, van Duijnhoven FJ, Kampman E. The COLON study: Colorectal cancer: Longitudinal, Observational study on Nutritional and lifestyle factors that may influence colorectal tumour recurrence, survival and quality of life. BMC Cancer. 2014 May 27;14:374. doi: 10.1186/1471-2407-14-374. PMID 24886284
- [Background] Veettil SK, Wong TY, Loo YS, Playdon MC, Lai NM, Giovannucci EL, Chaiyakunapruk N. Role of Diet in Colorectal Cancer Incidence: Umbrella Review of Meta-analyses of Prospective Observational Studies. JAMA Netw Open. 2021 Feb 1;4(2):e2037341. doi: 10.1001/jamanetworkopen.2020.37341. PMID 33591366
- [Background] Njor SH, Andersen B, Friis-Hansen L, de Haas N, Linnemann D, Norgaard H, Roikjaer O, Sondergaard B, Rasmussen M. The optimal cut-off value in fit-based colorectal cancer screening: An observational study. Cancer Med. 2021 Mar;10(5):1872-1879. doi: 10.1002/cam4.3761. Epub 2021 Feb 3. PMID 33534955

DOCUMENTS (1):
  • Informed Consent Form (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT05891730/ICF_000.pdf